CLINICAL TRIAL: NCT05232812
Title: Human Ketone Metabolism - Validation of 3-[11C]-OHB as a New PET Ketontracer
Brief Title: Validation of 3-[11C]-OHB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1-10-72-290-20
Record Dates: First submitted 2022-01-10; First posted 2022-02-10 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 2; Heart Failure; Healthy
Keywords: Ketone bodies; Whole-body biodistribution
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of 3-[11C]-OHB (Experimental): All participants will first be injected with 200 MBq 3-[11C]-OHB followed by an oral ingestion of 100 MBq 3-[11C]-OHB.
  Interventions: Radiation: 3-[11C]-OHB

INTERVENTIONS:
Radiation: 3-[11C]-OHB — The PET tracer 3-[11C]-OHB is used to quantify 3-hydroxybutyrate uptake

SUMMARY:
Ketone bodies are produced in the liver at high levels of fatty acids, and act as an important source of energy for the brain and heart during fasting. The energy production from ketone metabolism is less oxygen-demanding than both glucose and fatty acid metabolism, and ketone substances can therefore be a very energy-efficient substrate for the heart. Insulin-resistant people as well as people with heart disease have difficulty burning glucose in the heart due to the insulin resistant condition and are therefore dependent on other energy sources such as free fatty acids and ketones. Because ketones are oxygen-sparing compared to fatty acids, interventions that increase the level of ketone bodies can potentially reduce the heart's need for oxygen in patients with narrowed coronary arteries. PET/CT is a functional and non-invasive imaging modality and suitable for tracking the fate of metabolites non-invasively, as most substrates or metabolites can be labeled by a PET isotope.

The purpose of this experiment is therefore to validate a new ketone tracer called 3-[11C]-OHB. Implementation of the 3-[11C]-OHB tracer will in future allow the investigators to more directly estimate the impact of different levels of ketone bodies on organ functions by measuring tissue-specific ketone uptake, both after intravenous and oral administration.

DETAILED DESCRIPTION:
Background:

Ketone bodies consists of 3-hydroxybutyrat, acetoacetate, and acetone. They are produced in the liver at high levels of fatty acids, and act as an important source of energy for the heart, brain and skeletal muscle during fasting. Energy production by ketone metabolism is less oxygen-intensive than both glucose and fatty acid metabolism, and ketone substances can therefore be a highly energy-efficient substrate. Insulin resistant individuals as well as people with heart disease have difficulty utilising glucose in the heart due to the insulin resistant condition and are therefore dependent on other energy sources such as free fatty acids and ketones. Because ketones are oxygen sparing compared to fatty acids, interventions that increase the level of ketone bodies can potentially reduce the heart's need for oxygen in patients with narrowed coronary arteries. This has led to an increased focus on the potential of ketone bodies in the treatment of a number of diseases, including especially cardiovascular disease.

Our group has shown that ketone bodies are efficiently absorbed by the heart despite maximal stimulation with insulin and glucose. In the study, healthy subjects increased the level of circulating ketone bodies to approximately 4 millimolar with a continuous ketone infusion, which resulted in a 50% reduction in cardiac glucose consumption. Since the consumption of free fatty acids in the experiment was unchanged and the overall work of the heart was the same, up to 50% of the heart's energy consumption was thus covered by ketone bodies. In addition, the high levels of ketone bodies led to a marked increase in the blood flow to the heart, which could potentially further benefit patients with narrowed coronary arteries

PET/CT is a functional and non-invasive imaging modality that is well established in oncological staging and treatment monitoring. The technique is also suitable for tracking the fate of metabolites non-invasively, as most substrates or metabolites can be labeled by a suitable PET isotope. PET has sufficient spatial and temporal resolution to enable direct quantification of e.g. uptake and oxidation rates and has been successfully used by our department to assess heart efficiency, oxygen consumption and fatty acid metabolism.

Purpose With this study, the investigators want to determine the metabolism of ketone bodies in healthy individuals and validate a newly developed ketone PET tracer for use in humans called 3-[11C]-OHB. Previous studies conducted by our and others' groups have only been able to indirectly estimate the uptake of ketone bodies into the heart. With 3-[11C]-OHB, the investigators will be able to directly measure tissue-specific ketone uptake, both after intravenous and oral administration.

Ihe investigators will apply state-of-the-science PET/CT tracer techniques and well-established models for estimating ketone metabolism (kinetics) and the radiation exposure of the tracer. Implementation of the 11C-3-OHB tracer in the future will allow the investigators to more directly estimate the impact of different levels of ketone bodies on organ functions, not least in the heart.

In this study, the investigators plan specifically

* To investigate the biodistribution and kinetics of the tracer 3-[11C]-OHB
* To estimate the radiation exposure of 3-[11C]-OHB by intravenous and oral administration of the tracer

Methods:

Six healthy and overweight (BMI: 28-40 kg/m^2) aged 50-70 years will undergo two PET/CT scans with 3-[11C]-OHB. One scan will be performed with the injection of 200 MBq of tracer and the other one will be performed with the subjects orally ingestion 100 MBq of the tracer. Following administration of the tracer, dynamic PET scans over the whole body will be performed to measure the biodistribution and radiation exposure of the tracer.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50-70 years
* BMI: 20-30 kg/m^2

Exclusion Criteria:

* All drugs that could affect the outcome
* HbA1c > 48 mmol/mol
* Known heart failure og episodes of acute myocardial infarction
* Liver disease ALAT > higher than 3 times of the normal level
* Kidney disease eGFR < 60 ml/min
* Blood donation in the last 3 months before inclusion
* Participation in other studies with radiation in the last 6 months
* Alcohol addiction

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Biodistribution of 3-[11C]-OHB | Through study completion, an average of 6 months
  The investigators will measure time activity curves by quantifying uptake of the PET ketone tracer 3-[11C]-OHB in kilo becquerel/ml over time (seconds).
Radiation exposure of 3-[11C]-OHB | Through study completion, an average of 6 months
  The investigators will measure radiation exposure of 3-[11C]-OHB in millisievert in relevant organs.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Jutland, Denmark

REFERENCES:
- [Derived] Luong TV, Nielsen EN, Falborg L, Kjaerulff MLG, Tolbod LP, Sondergaard E, Moller N, Munk OL, Gormsen LC. Intravenous and oral whole body ketone dosimetry, biodistribution, metabolite correction and kinetics studied by (R)-[1-11C]beta-hydroxybutyrate ([11C]OHB) PET in healthy humans. EJNMMI Radiopharm Chem. 2023 Jun 14;8(1):12. doi: 10.1186/s41181-023-00198-z. PMID 37314530